CLINICAL TRIAL: NCT05059405
Title: Pashto Translation, Validity and Reliability of Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale in Spinal Cord Injuries
Brief Title: Pashto Translation of Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC01035 Habib Khan
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injuries
Keywords: Pain
MeSH Terms: conditions — Spinal Cord Injuries; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a need for a culturally adapted screening tool to aid health care professionals or clinicians screen for the presence of neuropathic pain associated with spinal cord injuries in Pashtoon population. . Since Paraplegic center Hayatabad Peshawar is a reputable institute for spinal cord injury patients' rehabilitation in Khyber pakhtun khwa where most of Pashto speaking SCI patients are rehabilitated. While working there as a physical therapist I, my other colleagues and patients felt a need for a screening tool for pain in Pashto language .So I decided to a conduct a tool validation study. This study will help the clinicians to assess their patient's pain type easily through the Pashto version of LANSS pain scale in Pashtoon population and hence will help in timely management of the pain.

DETAILED DESCRIPTION:
The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale, a screening questionnaire for identifying patients with neuropathic pain, was developed to identify patients with neuropathic mechanisms dominating their pain experience. The original English version of the LANSS pain scale has been translated and validated in Turkish, Spanish, Swedish, Brazilian, Portuguese, and Chinese Mandarin languages. However, no neuropathic pain questionnaire including the LANSS has yet been established in Pasto language in Pakistan.

Although these screening tools are based on descriptors, their linguistic adaptation and validation into different languages are feasible and this ensures their reliability and validity in languages other than those in which they were initially developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic spinal cord injury
* Both Complete and Incomplete SCI patients
* Patients having pain history after spinal cord injury
* Patients having 3 or more than 3 months duration of SCI
* SCI at or below thoracic spine

Exclusion Criteria:

* Patients with other neurological disorders like multiple sclerosis, GBS, etc.
* Congenital conditions, tumor etc.
* Diabetic patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: spinal cord injury patients
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Pashto version of Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale | 1 week
  Pashto version of the LANSS will be developed through our study which will be same in contents to English version and will be applied on the spinal cord injury patients for validity and reliability in Pashtoon population.
Douleur Neuropathique 4 Questions (DN4) questionnaire | 1 week
  The DN4 questionnaire consists of a total of 10 items grouped in 4 sections . The first seven items are related to the quality of pain (burning, painful cold, electric shocks) and its association to abnormal sensations (tingling, pins and needles, numbness, itching). The other 3 items are related to neurological examination in the painful area (touch hypoesthesia, pinprick hypoesthesia, tactile allodynia). A score of 1 is given to each positive item and a score of 0 to each negative item. The total score is calculated as the sum of all 10 items, and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Paraplegic Center, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No